CLINICAL TRIAL: NCT02351752
Title: Renal Division, Peking University First Hospital, Institute of Nephrology, Peking University, Key Laboratory of Renal Disease
Brief Title: Hydroxychloroquine Sulfate for Reduction of Proteinuria in Patients With IgA Nephropathy: a Self- Controlled Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LLiu (Other)
Responsible Party: Sponsor-Investigator, LLiu, Renal Division, Peking University First Hospital, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014【851】
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxychloroquine Sulfate (Experimental): Hydroxychloroquine Sulfate 0.1 Tid (eGFR 30-59), 0.2 Bid(eGFR >60)
  Interventions: Drug: Hydroxychloroquine Sulfate

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — Hydroxychloroquine Sulfate: 0.1 Tid(eGFR 30-59);0.2 Bid (eGFR>60)

SUMMARY:
IgA nephropathy is the most common type of primary glomerulonephritis and might caused by deposition of immune complex containing IgA in mesangium and causing local immune activation. Hydroxychloroquine reduces the activation of dendritic cells and the inflammatory process and showed the potential effect of treatment of patients with IgA nephropathy.

The investigators study will recruite IgA nephropathy patients with proteinuria range from 0.75 to 3.5g/d even after three-month treatment by sufficient ACEi/ARB. The patients were treated with Hydroxychloroquine 300-400mg/d according to eGFR. The proteinuria will recorded every two months and total four months. Then, the drug will be stopped for two months for observation of change of proteinuria.

DETAILED DESCRIPTION:
Immunoglobulin A (IgA) nephropathy is the most common type of primary glomerulonephritis worldwide. Several studies indicated that 6-43% of IgA nephropathy patients would develop end-stage kidney disease (ESKD) over a period of 10 years. The clinical risk factors for progression are hypertension, protienuria, impaired renal function and histologic lesions at presentation. There is no well accepted optimal therapy for patients with IgA. Current established therapies include full RAS inhibition and optimal blood pressure control for patients with proteinuria and/or hypertension.

Hydroxychloroquine has been used for many years to treat malaria. It is also used to treat systemic lupus erythematosus, rheumatic disorders like rheumatoid arthritis and Sjögren's Syndrome. Recently, several studies found that Hydroxychloroquine could reduce the risk of ESRD in patients with lupus nephrits. The mechanism of the treatment wasn't well known so far. Some investigators found that Hydroxychloroquine increases lysosomal pH in antigen presenting cells. In inflammatory conditions, it blocks toll-like receptors on plasmacytoid dendritic cells (PDCs). Toll-like receptor 9 (TLR 9), which recognizes DNA-containing immune complexes, leads to the production of interferon and causes the dendritic cells to mature and present antigen to T cells. Hydroxychloroquine, by decreasing TLR signaling, reduces the activation of dendritic cells and the inflammatory process.

The pathogenesis of IgA nephropathy included the deposition of immune complex containing IgA in mesangium and causing local immune activation and injury to kidney. Therefore, Hydroxychloroquine might have the potential effect of anti-inflammation in patients with IgA nephropathy, reduced the proteinuria and had the renal protect effect.

Our study will recruite IgA nephropathy patients with proteinuria range from 0.75 to 3.5g/d even after three-month treatment by sufficient ACEi/ARB. The patients were treated with Hydroxychloroquine 300-400mg/d according to eGFR. The proteinuria will recorded every two months and total four months. Then, the drug will be stopped for two months for observation of change of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

1. primary IgA nephopathy
2. age 18-75 years
3. proteinuria range from 0.75 to 3.5g/d even after three-month treatment by sufficient ACEi/ARB
4. eGFR>30ml/min/1.73m2

Exclusion Criteria:

1. immune suppressive agent in recent one years
2. crescent glomerulonephritis, might use immune suppressive agent
3. chronic hepatic disease
4. myocardial infarction
5. malignant hypertension
6. stroke
7. malignant tumor
8. retinopathy
9. other contraindication of Hydroxychloroquine
10. pregnancy and breastfeeding women
11. life expectancy for less than 6 months
12. in other clinical trials
13. not suitable for the study judged by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
proteinuia | total four months(proteinic will recorded every 2 months )

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, PhD,MD, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China